CLINICAL TRIAL: NCT06178120
Title: An Observational Study to Assess Disease Progression in Women With X-linked Adrenoleukodystrophy
Brief Title: Disease Progression in Women With X-linked Adrenoleukodystrophy
Status: Recruiting | Type: Observational
Sponsor: Minoryx Therapeutics, S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: MT-NH-01
Record Dates: First submitted 2023-11-28; First posted 2023-12-20 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-12

CONDITIONS: X-linked Adrenoleukodystrophy
MeSH Terms: conditions — Adrenoleukodystrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational, single-site prospective and minimally interventional study in women with X-linked adrenoleukodystrophy (ALD), conducted in France.

DETAILED DESCRIPTION:
Patients accepting participation (after signing ICF) will be followed up to at least 2 years or until they started treatment for X-linked adrenoleukodystrophy (ALD) or withdraw consent, whichever occurs first. Follow-up will be extended beyond 2 years if deemed appropriate after an interim report. Tests and questionnaires will be assessed at baseline and yearly. If the study is extended, beyond 2 years, patients will be assessed at 1-year intervals.

At baseline visit and follow-up visits, patients will undergo an MRI of the brain and the spinal cord and assessments of body sway, EDSS, ADL, pain VAS and SF-36 questionnaire. Plasma biomarkers will be assessed from samples obtained through routine blood draw and a monthly falls diary will be provided each visit to be completed once a month.

This study will not assess any specific medicinal product or intervention, and the study will not interfere with that prescribed in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 years old or older.
2. Diagnosis of X-linked ALD based on genetic testing, altered VLCFA levels, or family history.
3. Willing to undergo annual follow-up visits, including brain and spinal cord MRI scans.
4. Provision of written informed consent.
5. Affiliation or beneficiary of a French social security system or of such a regime.

Exclusion Criteria:

1. Any condition that in the opinion of the investigator are likely to adversely affect the study participation, interfere with study compliance, or confound the study results.
2. Under treatment or previous treatment with leriglitazone.
3. Pregnant or lactating women.
4. Subjects benefiting from laws aimed at protecting vulnerable adults: subjects being deprived of liberty by judicial or administrative decision, subjects under guardianship.
5. Participation in an interventional clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include up to 40 adult women with X-linked ALD who attend to a regular visit, who meet all inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Spinal cord magnetization transfer ratio (MTR) | Change from baseline up to 2 years
  To assess the disease evolution on spinal cord MRI

SECONDARY OUTCOMES:
Spinal cord morphometry. Cross sectional area (CSA) to cover the C1 to C7 vertebral levels. | Change from baseline up to 2 years
  To assess the disease evolution on spinal cord MRI
Spinal cord diffusion image analysis parameters: Fractional Anisotropy (FA), Radial Diffusivity (RD), Axial Diffusivity (AD), Mean Diffusivity (MD) at the cervical levels C1-C5. | Change from baseline up to 2 years
  To assess the disease evolution on spinal cord MRI
Brain diffusion image analysis parameters: Fixel-Based analysis (FBA) (Fiber Density (FD), Fiber cross-section (FC) and combination of FD and FC), Diffusion tensor imaging (DTI) (FA, RD, AD, MD, Markers of severity and markers of evolution). | Change from baseline up to 2 years
  To assess the disease evolution on brain MRI
Body sway amplitude (considering antero-posterior and medio-lateral sway with eyes closed, feet apart; eyes open, feet apart; eyes closed, feet together; eyes open, feet together) | Change from baseline up to 2 years
  To assess clinical evolution of myelopathy
Expanded Disability Status Scale (EDSS) | Change from baseline up to 2 years
  To assess the impact on Quality of Life
Activities of Daily Living (ADL) | Change from baseline up to 2 years
  To assess the impact on Quality of Life
Pain Visual Analogue Scale (Pain VAS) | Change from baseline up to 2 years
  To assess the impact on Quality of Life
Monthly falls | Change from baseline up to 2 years
  To assess the impact on Quality of Life
Short Form Health Survey (SF-36) | Change from baseline up to 2 years
  To assess the impact on Quality of Life
Plasma biomarkers (NFL, MMP-9, IL-18, MIP-1beta and IL-1Ra) | Change from baseline up to 2 years
  To assess the evolution of plasma biomarkers

CONTACTS AND LOCATIONS:
Locations (1):
- Paris Brain Institute (ICM) Centre Hospitalier Universitaire Pitié Salpêtrière, Paris, France